CLINICAL TRIAL: NCT03408470
Title: A 2-Cohort Study to Evaluate the Absolute Bioavailability, Absorption, Distribution, Metabolism and Excretion of TD-1473 Following an Intravenous and an Oral Dose of [14C]-TD-1473 in Healthy Male Subjects
Brief Title: TD-1473 Absorption, Distribution, Metabolism and Excretion (ADME) Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0152
Record Dates: First submitted 2018-01-12; First posted 2018-01-24 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Intestinal Disorders; Bowel Diseases, Inflammatory
Keywords: Absolute Bioavailability; ADME; Healthy Normal Males
MeSH Terms: conditions — Intestinal Diseases; Inflammatory Bowel Diseases | interventions — izencitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TD-1473 Oral Capsule & [14C]-TD-1473 IV bolus (Experimental): Cohort 1 - One oral dose and IV bolus administered 1 hr after oral dose of TD-1473
  Interventions: Drug: TD-1473 oral capsule; Drug: [14C]-TD-1473 IV bolus
- [14C]-TD-1473 Oral Capsule (Experimental): Cohort 2 - One oral dose
  Interventions: Drug: [14C]-TD-1473 Oral Capsule

INTERVENTIONS:
Drug: TD-1473 oral capsule — (Intervention description included in arm description)
  Arms: TD-1473 Oral Capsule & [14C]-TD-1473 IV bolus
Drug: [14C]-TD-1473 IV bolus — (Intervention description included in arm description)
  Arms: TD-1473 Oral Capsule & [14C]-TD-1473 IV bolus
Drug: [14C]-TD-1473 Oral Capsule — (Intervention description included in arm description)
  Arms: [14C]-TD-1473 Oral Capsule

SUMMARY:
This is an open-label, 2-cohort study to evaluate the absolute bioavailability, absorption, distribution, metabolism and excretion of TD-1473 in healthy male subjects. Subjects in cohort 1 will receive a single oral dose of TD-1473 and a single intravenous bolus dose of [14C]-TD-1473. Subjects in cohort 2 will receive a single oral dose of [14C]-TD-1473 only.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy, nonsmoking male, 19 to 55 years old, inclusive
* Subject has a body mass index (BMI) 19 to 32 kg/m2, inclusive, and weighs at least 50 kg
* Subject is healthy as determined by the PI or designee based on medical history and physical examination performed at Screening and Day -1
* Additional inclusion criteria apply

Exclusion Criteria:

* Subject has any condition possibly affecting drug absorption (e.g., previous surgery on the gastrointestinal tract [including removal of parts of the stomach, bowel, liver, gall bladder, or pancreas])
* Subject has a known hypersensitivity towards medications similar to TD 1473 or excipients contained in TD 1473
* Subject regularly works with ionizing radiation or radioactive material
* Subject has been exposed to ionizing radiations, within 1 year prior to the start of the study, as external irradiation (i.e., radiological examination including CT scan, excluding dental radiography) or internal radiation (i.e., diagnostic nuclear medicine procedure) or have participated in a radiolabeled study in the last 12 months
* Subject, who, for any reason, is deemed by the PI or designee or Sponsor to be inappropriate for this study or have any condition which would confound or interfere with the evaluation of the safety, tolerability, and PK of the investigational drug or prevent compliance with the study protocol
* Additional exclusion criteria apply

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males only
Enrollment: 20 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) in Plasma | Up to 15 days
Time to maximum observed concentration (tmax) in Plasma | Up to 15 days
Area under the concentration-time curve from hour 0 to the last measurable concentration (AUC0-last) in Plasma | Up to 15 days
Area under the concentration-time curve extrapolated to infinity (AUC0-inf) in Plasma | Up to 15 days
Apparent terminal elimination half-life (t1/2) in Plasma | Up to 15 days
Apparent clearance (Cl/F) in Plasma | Up to 15 days
Apparent volume of distribution (Vz/F) in Plasma | Up to 15 days
Absolute bioavailability (%F) in Plasma | Up to 15 days

SECONDARY OUTCOMES:
Amount excreted in urine (Aeu) over the sampling interval in Urine | Up to 15 days
Renal clearance (CLr) in Urine | Up to 15 days
The percent excreted in urine (%Feu) in Urine | Up to 15 days
Amount excreted in feces (Aef) over the sampling interval in Feces | Up to 15 days
The percent excreted in feces (%Fef) | Up to 15 days

OTHER OUTCOMES:
Metabolites in Plasma | Up to 15 days
  TD 1473 metabolite profiling will be performed in plasma containing sufficient amounts of radioactivity
Metabolites in Urine | Up to 15 days
  TD 1473 metabolite profiling will be performed in urine containing sufficient amounts of radioactivity
Metabolites in Feces | Up to 15 days
  TD-1473 metabolite profiling will be performed in feces containing sufficient amounts of radioactivity

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Theravance Biopharma, Inc. will not be sharing individual de-identified participant data or other relevant study documents.